CLINICAL TRIAL: NCT04579250
Title: VRC 323: A Phase I Open-Label Clinical Trial to Evaluate the Dose, Safety, Tolerability and Immunogenicity of an Influenza H10 Stabilized Stem Ferritin Vaccine, VRC-FLUNPF0103-00-VP, in Healthy Adults
Brief Title: Dose, Safety, Tolerability and Immunogenicity of an Influenza H10 Stabilized Stem Ferritin Vaccine, VRC-FLUNPF0103-00-VP, in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 200145; 20-I-0145 (Other: NIH IRB)
Record Dates: First submitted 2020-10-07; First posted 2020-10-08 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Influenza
Keywords: Flu Virus; Respiratory Illness; Viral Infection; Experimental Vaccine
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: H10ssF-6473 (20 mcg), ages 18-50 years (Experimental): H10ssF-6473 (20 mcg) administered intramuscularly (IM) by Needle/Syringe (Day 0)
  Interventions: Biological: VRC-FLUNPF0103-00-VP (H10ssF-6473)
- Group 2A: H10ssF-6473 (60 mcg), ages 18-50 years (Experimental): H10ssF-6473 (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16)
  Interventions: Biological: VRC-FLUNPF0103-00-VP (H10ssF-6473)
- Group 2B: H10ssF-6473 (60 mcg), ages 55-70 years (Experimental): H10ssF-6473 (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16)
  Interventions: Biological: VRC-FLUNPF0103-00-VP (H10ssF-6473)

INTERVENTIONS:
Biological: VRC-FLUNPF0103-00-VP (H10ssF-6473) — The vaccine is composed of the haemagglutinin (HA) stem domain from A/Jiangxi/IPB13/2013 (H10N8) influenza genetically fused to the ferritin protein from H. pylori. Purified H10ssF-6473 displays eight well-formed HA trimers that antigenically resemble the native H10 stem viral spikes.

SUMMARY:
Background: The flu is a common viral infection that can be deadly for certain people. Vaccines against flu have been developed to teach the body to prevent or fight the infection. A new vaccine may help the body to make an immune response to H10 flu, a flu strain that infects humans.

Objective:

To test the safety and effectiveness of the H10 Stabilized Stem Ferritin vaccine (VRC-FLUNPF0103-00-VP or H10ssF-6473).

Eligibility:

Healthy adults ages 18-70, but not born between 1965-1970

Design:

Participants received 1 or 2 vaccinations by injections (shots) in the upper arm muscle over 4 months. Participants received a thermometer and recorded their temperature and symptoms every day on/with/via a diary card for 7 days after each injection. The injection site was checked for redness, swelling, itching or bruising.

Participants had 8-10 follow-up visits over 10 months. At follow-up visits, participants had blood drawn and were checked for health changes or problems. Participants who reported influenza-like illness had nose and throat swabs collected for evaluation of viral infection.

Some participants had apheresis. A needle was placed into a vein in both arms. Blood was removed through a needle in the vein of one arm. A machine removed the white blood cells and then the rest of the blood was returned to the participant through a needle in the other arm.

DETAILED DESCRIPTION:
Design: This was a Phase I, open-label, dose escalation study to evaluate the dose, safety, tolerability, and immunogenicity of VRC-FLUNPF0103-00-VP in two regimens. The hypotheses were that the vaccine is safe and tolerable and would elicit an immune response. The primary objective was to evaluate the safety and tolerability of the investigational vaccine in healthy adults. Secondary objectives were related to immunogenicity of the investigational vaccine and dosing regimen.

Study Products: The investigational vaccine, VRC-FLUNPF0103-00-VP (H10ssF-6473), was developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Diseases (NIAID) and is composed of the haemagglutinin (HA) stem domain from A/Jiangxi/IPB13/2013 (H10N8) influenza genetically fused to the ferritin protein from Helicobacter pylori. Purified H10ssF-6473 displays eight well-formed HA trimers that antigenically resemble the native H10 stem viral spikes. The vaccine was supplied in single-use vials at a concentration of 180 mcg/mL. VRC-PBSPLA043-00-VP consisting of sterile phosphate buffered saline (PBS) was the diluent for H10ssF-6473. Prepared study product was administered intramuscularly (IM) in the deltoid muscle via needle and syringe.

Participants:

Healthy adults between the ages of 18-70 were enrolled; adults born between 1965 and 1970 were excluded from the trial

Study Plan: This study evaluated the safety, tolerability and immunogenicity of 1 or 2 doses of H10ssF-6473 in a dose-escalation design.

In Group 1, three participants received a single low dose (20 mcg) of H10ssF-6473 on Day 0. For Group 1, the protocol required 1 vaccination visit, 8 follow-up visits, and a telephone contact after vaccination.

Once the low dose was assessed as safe and well tolerated, enrollment began for Group 2A. In Group 2A, participants received a higher dose (60 mcg) of H10ssF-6473 on Day 0. Once this higher dose was assessed as safe and well tolerated, participants in Group 2A received a second vaccination at Week 16 and enrollment began for Groups 2B. Groups 2A and 2B were stratified by age as shown in the vaccination schema below. For Groups 2A and 2B, the protocol required 2 vaccination visits, 10 follow-up visits, and a telephone contact after each vaccination.

For all groups, solicited reactogenicity was evaluated using a 7-day diary card. Assessment of vaccine safety included clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

VRC 323 Vaccination Schema:

Group: 1; Age Cohort: 18-50; Participants: 3; Day 0: 20 mcg IM

Group: 2A; Age Cohort: 18-50; Participants: 14; Day 0: 60 mcg IM, Week 16: 60 mcg IM

Group: 2B; Age Cohort: 55-70; Participants: 8; Day 0: 60 mcg IM, Week 16: 60 mcg IM

Total Participants: 25

Study Duration:

Participants were evaluated for 40 weeks following the first vaccine administration.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Healthy adults between the ages of 18-70 years (excluding adults born between January 1, 1965 and December 31,1970)
2. Based on history and examination, in good general health and without history of any of the conditions listed in the exclusion criteria
3. Received at least one licensed influenza vaccine from 2015 to the present
4. Able and willing to complete the informed consent process
5. Available for clinic visits for 40 weeks after enrollment
6. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
7. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than or equal to 40 within the 56 days before enrollment

   Laboratory Criteria within 56 days before enrollment
8. White blood cells (WBC) and differential within institutional normal range or accompanied by the site Principal Investigator (PI) or designee approval
9. Total lymphocyte count greater than or equal to 800 cells/microL
10. Platelets = 125,000 - 500,000 cells/microL
11. Hemoglobin within institutional normal range or accompanied by the PI or designee approval
12. Serum iron within institutional normal range or accompanied by the site PI or designee approval
13. Serum ferritin within institutional normal range or accompanied by the site PI or designee approval
14. Alanine aminotransferase (ALT) less than or equal to 1.25 x institutional upper limit of normal (ULN)
15. Aspartate aminotransferase (AST) less than or equal to 1.25 x institutional ULN
16. Alkaline phosphatase (ALP) <1.1 x institutional ULN
17. Total bilirubin within institutional normal range, except when otherwise consistent with Gilbert's syndrome
18. Serum creatinine less than or equal to 1.1 x institutional ULN
19. Negative for HIV infection by an FDA-approved method of detection

    Criteria applicable to women of childbearing potential:
20. Negative beta-human chorionic gonadotropin (Beta-HCG) pregnancy test (urine or serum) on the day of enrollment
21. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through the end of the study

EXCLUSION CRITERIA:

1. Breast-feeding or planning to become pregnant during the study

   Individual has received any of the following substances:
2. More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
3. Blood products within 16 weeks prior to enrollment
4. Live attenuated vaccines within 4 weeks prior to enrollment
5. Inactivated vaccines within 2 weeks prior to enrollment
6. Investigational research agents within 4 weeks prior to enrollment or planning to receive investigational products while on the study
7. Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule
8. Current anti-TB (tuberculosis) prophylaxis or therapy
9. Previous investigational H10 influenza vaccine
10. Receipt of a licensed influenza vaccine within 6 weeks prior to enrollment

    Individual has a history of any of the following clinically significant conditions:
11. Serious reactions to vaccines that preclude receipt of the study vaccination as determined by the investigator
12. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
13. Asthma that is not well controlled
14. Diabetes mellitus (type I or II), with the exception of gestational diabetes
15. Thyroid disease that is not well controlled
16. Idiopathic urticaria within the past year
17. Autoimmune disease or immunodeficiency
18. Hypertension that is not well controlled (baseline systolic > 140 mmHg or diastolic > 90 mmHg)
19. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
20. Malignancy that is active or history of malignancy that is likely to recur during the period of the study
21. Seizure disorder other than 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
22. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
23. Guillain-Barre Syndrome
24. Previous or current infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) documented by polymerase chain reaction (PCR) test
25. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant's ability to give informed consent.

INCLUSION OF VULNERABLE PARTICIPANTS

Children

Children were not eligible to participate in this clinical trial because the investigational vaccine had not been previously evaluated in adults. If the product is assessed as safe and immunogenic, other protocols designed for children may be conducted in the future.

NIH Employees

NIH employees and members of their immediate families could have participated in this protocol. If eligible, the Guidelines for the Inclusion of Employees in NIH Research Studies were followed for employees and each employee was given a copy of the 'NIH Information Sheet on Employee Research Participation' and a copy of the 'Leave Policy for NIH Employees Participating in NIH Medical Research Studies.'

Neither participation nor refusal to participate had an effect, either beneficial or adverse, on the participant's employment or work situation. The NIH information sheet regarding NIH employee research participation was distributed to all potential participants who are NIH employees. The employee participant's privacy and confidentiality was preserved in accordance with NIH Clinical Center and NIAID policies. For NIH employee participants, consent was obtained by an individual who is independent of the participant's team. If the individual obtaining consent is a co-worker to the participant, independent monitoring of the consent process will be included through the Bioethics Consultation Service. Protocol study staff were trained on obtaining potentially sensitive and private information from co-workers or subordinates.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Casazza, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledgerwood JE, Zephir K, Hu Z, Wei CJ, Chang L, Enama ME, Hendel CS, Sitar S, Bailer RT, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 310 Study Team. Prime-boost interval matters: a randomized phase 1 study to identify the minimum interval necessary to observe the H5 DNA influenza vaccine priming effect. J Infect Dis. 2013 Aug 1;208(3):418-22. doi: 10.1093/infdis/jit180. Epub 2013 Apr 30. PMID 23633407
- [Background] Kanekiyo M, Wei CJ, Yassine HM, McTamney PM, Boyington JC, Whittle JR, Rao SS, Kong WP, Wang L, Nabel GJ. Self-assembling influenza nanoparticle vaccines elicit broadly neutralizing H1N1 antibodies. Nature. 2013 Jul 4;499(7456):102-6. doi: 10.1038/nature12202. Epub 2013 May 22. PMID 23698367
- [Background] Boyoglu-Barnum S, Hutchinson GB, Boyington JC, Moin SM, Gillespie RA, Tsybovsky Y, Stephens T, Vaile JR, Lederhofer J, Corbett KS, Fisher BE, Yassine HM, Andrews SF, Crank MC, McDermott AB, Mascola JR, Graham BS, Kanekiyo M. Glycan repositioning of influenza hemagglutinin stem facilitates the elicitation of protective cross-group antibody responses. Nat Commun. 2020 Feb 7;11(1):791. doi: 10.1038/s41467-020-14579-4. PMID 32034141
- [Background] Houser KV, Chen GL, Carter C, Crank MC, Nguyen TA, Burgos Florez MC, Berkowitz NM, Mendoza F, Hendel CS, Gordon IJ, Coates EE, Vazquez S, Stein J, Case CL, Lawlor H, Carlton K, Gaudinski MR, Strom L, Hofstetter AR, Liang CJ, Narpala S, Hatcher C, Gillespie RA, Creanga A, Kanekiyo M, Raab JE, Andrews SF, Zhang Y, Yang ES, Wang L, Leung K, Kong WP, Freyn AW, Nachbagauer R, Palese P, Bailer RT, McDermott AB, Koup RA, Gall JG, Arnold F, Mascola JR, Graham BS, Ledgerwood JE; VRC 316 Study Team. Safety and immunogenicity of a ferritin nanoparticle H2 influenza vaccine in healthy adults: a phase 1 trial. Nat Med. 2022 Feb;28(2):383-391. doi: 10.1038/s41591-021-01660-8. Epub 2022 Feb 3. PMID 35115706
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0145.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the NIH Clinical Center in Bethesda, Maryland.
Period: Overall Study
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years
Started | 3 | 14 | 8
Received First Product Administration | 3 | 14 | 8
Completed Product Administrations | 3 | 14 | 8
Completed | 1 | 11 | 6
Not Completed | 2 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Moved from area | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Total
Number analyzed (Participants) | 3 | 14 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (7.6) | 29.9 (8.2) | 60.5 (4.2) | 40.2 (15.8)
Age, Customized [Count of Participants; unit: Participants]
  21-30 years | 1 | 7 | 0 | 8
  31-40 years | 1 | 5 | 0 | 6
  41-50 years | 1 | 2 | 0 | 3
  51-60 years | 0 | 0 | 4 | 4
  61-70 years | 0 | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 3 | 10
  Male | 2 | 8 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 2 | 6
  Not Hispanic or Latino | 3 | 10 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 2 | 6 | 6 | 14
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (2.9) | 26.2 (4.0) | 28.7 (3.4) | 27.0 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Each H10ssF-6473 Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after each H10ssF-6473 product administration, at approximately Week 1 and at approximately Week 17
Population: Population included all enrolled participants who received at least one H10ssF-6473 study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=25).
Measure: Count of Participants; unit: Participants
Groups:
- Overall Incidence H10ssF-6473 (20 mcg and 60 mcg): H10ssF-6473 dose groups included adults who received at least one dose of H10ssF-6473.
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Incidence H10ssF-6473 (20 mcg and 60 mcg)
Number analyzed (Participants) | 3 | 14 | 8 | 25
Participants
  Pain/Tenderness: None | 3 | 9 | 5 | 17
  Pain/Tenderness: Mild | 0 | 5 | 3 | 8
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0
  Swelling: None | 3 | 14 | 7 | 24
  Swelling: Mild | 0 | 0 | 1 | 1
  Swelling: Moderate | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0
  Redness: None | 3 | 14 | 8 | 25
  Redness: Mild | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0
  Pruritis (Itching): None | 3 | 14 | 8 | 25
  Pruritis (Itching): Mild | 0 | 0 | 0 | 0
  Pruritis (Itching): Moderate | 0 | 0 | 0 | 0
  Pruritis (Itching): Severe | 0 | 0 | 0 | 0
  Bruising: None | 3 | 14 | 8 | 25
  Bruising: Mild | 0 | 0 | 0 | 0
  Bruising: Moderate | 0 | 0 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0
  Any Local Symptom: None | 3 | 9 | 5 | 17
  Any Local Symptom: Mild | 0 | 5 | 3 | 8
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Each H10ssF-6473 Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after each H10ssF-6473 product administration, at approximately Week 1 and at approximately Week 17
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Incidence H10ssF-6473 (20 mcg and 60 mcg)
Number analyzed (Participants) | 3 | 14 | 8 | 25
Participants
  Malaise: None | 2 | 9 | 8 | 19
  Malaise: Mild | 1 | 5 | 0 | 6
  Malaise: Moderate | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0
  Myalgia: None | 3 | 11 | 7 | 21
  Myalgia: Mild | 0 | 3 | 1 | 4
  Myalgia: Moderate | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0
  Headache: None | 3 | 13 | 6 | 22
  Headache: Mild | 0 | 1 | 2 | 3
  Headache: Moderate | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0
  Chills: None | 3 | 12 | 8 | 23
  Chills: Mild | 0 | 2 | 0 | 2
  Chills: Moderate | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0
  Nausea: None | 3 | 14 | 7 | 24
  Nausea: Mild | 0 | 0 | 1 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0
  Temperature (Fever): None | 3 | 14 | 8 | 25
  Temperature (Fever): Mild | 0 | 0 | 0 | 0
  Temperature (Fever): Moderate | 0 | 0 | 0 | 0
  Temperature (Fever): Severe | 0 | 0 | 0 | 0
  Joint Pain: None | 3 | 13 | 8 | 24
  Joint Pain: Mild | 0 | 1 | 0 | 1
  Joint Pain: Moderate | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 2 | 7 | 6 | 15
  Any Systemic Symptom: Mild | 1 | 7 | 2 | 10
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following H10ssF-6473 Product Administration
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of the first study product administration through the visit scheduled for 4 weeks after each study product administration. At other time periods between study product administrations and when greater than 4 weeks after the last study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module), influenza-like illness (ILI) or influenza and new chronic medical conditions that required ongoing medical management (reported as separate outcomes) were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks after each H10ssF-6473 product administration, up to Week 20
Population: Population included all enrolled participants who received at least one H10ssF-6473 study injection (N=25).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Incidence H10ssF-6473 (20 mcg and 60 mcg)
Number analyzed (Participants) | 3 | 14 | 8 | 25
Participants
  Related to Study Product | 1 | 4 | 0 | 5
  Unrelated to Study Product | 1 | 7 | 5 | 13
  Total Number of Participants who had One or More Non-Serious Unsolicited AE | 2 | 11 | 5 | 18

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following H10ssF-6473 Product Administration
Description: SAEs were recorded from receipt of first study product administration through the last expected study visit at Week 40. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after H10ssF-6473 product administration through the study participation, up to Week 40
Population: Population included all enrolled participants who received at least one H10ssF-6473 study injection (N=25).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Incidence H10ssF-6473 (20 mcg and 60 mcg)
Number analyzed (Participants) | 3 | 14 | 8 | 25
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Influenza or Influenza-like Illness (ILIs) Following H10ssF-6473 Product Administration
Description: Influenza or influenza-like illness (ILI) were recorded in the study database from receipt of the first study product administration through the last study visit. ILI was defined as fever (temperature of 100 degrees F [37.8 degrees C] or greater) and a cough and/or sore throat in the absence of a known cause other than influenza. Collection of nasopharyngeal swabs were used for laboratory confirmation of influenza by polymerase chain reaction (PCR) in participants who met criteria for ILI. Subsequently, results of any reported laboratory testing for identification of pathogens were included for cases meeting initial criteria for ILI. The severity of illness in participants with laboratory confirmed influenza illness were captured on a case report form rather than on an Adverse Event (AE) form.
Time Frame: Day 0 after H10ssF-6473 product administration through the study participation, up to Week 40
Population: Population included all enrolled participants who received at least one H10ssF-6473 study injection (N=25).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Incidence H10ssF-6473 (20 mcg and 60 mcg)
Number analyzed (Participants) | 3 | 14 | 8 | 25
Participants
  Reported Influenza-like Illness | 0 | 1 | 0 | 1
  Influenza confirmed by clinical test | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following H10ssF-6473 Product Administration
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of first study product administration through the last expected study visit at Week 40. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after H10ssF-6473 product administration through the study participation, up to Week 40
Population: Population included all enrolled participants who received at least one H10ssF-6473 study injection (N=25).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Incidence H10ssF-6473 (20 mcg and 60 mcg)
Number analyzed (Participants) | 3 | 14 | 8 | 25
Participants
  Related to Study Product | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 2 | 2
  Total Number of Participants with New Chronic Medical Conditions | 0 | 0 | 2 | 2

7. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following H10ssF-6473 Product Administration
Description: Abnormal lab results recorded as unsolicited adverse events (AEs) are summarized. Safety lab parameters included hematology (hemoglobin, hematocrit, platelets, and white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil percents/counts) and chemistry (alanine aminotransferase (ALT), alanine aspartate (AST), alkaline phosphate (ALP), creatinine and total bilirubin). Complete Blood Count (CBC) with differential, total bilirubin, AST, ALT, and ALP results were collected at Day 14, 28, and 280 (Group 1) or at Day 14, 28, 112, 140 and 280 (Groups 2A-2B). Iron and serum ferritin were collected at Day 28 (Group 1) or at Days 112 and 140 (Groups 2A-2B). Creatinine results were collected at Day 14 (Group 1) or at Days 14 and 140 (Groups 2A-2B). Institutional lab normal ranges as well as Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials FDA Guidance, September 2007 were used.
Time Frame: Day 0 after H10ssF-6473 product administration through the study participation, up to Week 40
Population: Population included all enrolled participants who had laboratory results available at any study visit post product administration. If several cases of the same type of abnormal lab value/AE were detected in a participant, the participant was counted one time at the highest severity.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Incidence H10ssF-6473 (20 mcg and 60 mcg)
Number analyzed (Participants) | 3 | 14 | 8 | 25
Participants
  AST | 0 | 2 | 0 | 2
  WBC Count | 1 | 1 | 0 | 2
  Hemoglobin | 0 | 4 | 0 | 4
  Neutrophil Count | 1 | 1 | 0 | 2
  Lymphocyte Count | 0 | 1 | 0 | 1
  Number of Participants with one or more Abnormal Laboratory Results AE Related to Study Product | 1 | 4 | 0 | 5
  Number of Participants with one or more Abnormal Laboratory Results AE Unrelated to Study Product | 0 | 4 | 0 | 4
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 1 | 8 | 0 | 9

8. Secondary Outcome: Stem-Specific Antibody Response to H10ssF-6473 Following the Completion of Each Vaccination Regimen
Description: Stem-specific H10ss antibody titers were measured by Electrochemiluminescence Assay (ECLIA) using a Meso Scale Discovery (MSD) platform. Serum samples collected at baseline and at 2 weeks after the single and/or last product administration were tested in the assay. Area under the curve (AUC) was calculated for each serum sample tested in the 8-fold serial dilutions. The AUC measurement is calculated for each single timepoint sample (baseline, week 2: 2 weeks after the single vaccination and week 18: 2 weeks after the final vaccination). The AUC is calculated with GraphPad Prism™ using the trapezoid rule from the raw sample response (ECL response) over an 8-fold dilution series (dilution factor) for each sample. Group geometric mean AUCs and 95% Confidence Intervals are reported.
Time Frame: Baseline to 2 weeks after the single or first injection, at Week 2 and from Week 16 to 2 weeks after the second injection, at Week 18
Population: Baseline and Week 2 analyses included all who received at least one H10ssF-6473 study injection for which samples were available (N=25). Week 18 analysis included all who received two H10ssF-6473 injections for which samples were available (N=22).
Measure: Geometric Mean (95% Confidence Interval); unit: AUC (ECL response units/Dilution Factor)
Groups:
- Overall Group 2: H10ssF-6473 (60 mcg): H10ssF-6473 (60 mcg) dose groups included adults stratified by age (ages 18-50 years and ages 55-70 years) who were randomized to receive two doses of 60 mcg H10ssF-6473 16 weeks apart.
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Group 2: H10ssF-6473 (60 mcg)
Number analyzed (Participants) | 3 | 14 | 8 | 22
AUC (ECL response units/Dilution Factor)
  Week 0 (Baseline, Pre-Administration) | 2726.67 [492.87 to 15084.65] | 2421.80 [1872.73 to 3131.85] | 4122.82 [2988.15 to 5688.34] | 2938.72 [2364.13 to 3652.97]
  Week 2 (14 Days After First Product Administration) | 4796.47 [705.49 to 32609.97] | 6899.17 [5321.75 to 8944.16] | 5622.02 [3523.29 to 8970.92] | 6404.25 [5155.20 to 7955.93]
  Week 18 (14 Days After Second Product Administration): number analyzed (Participants) | 0 | 14 | 8 | 22
  Week 18 (14 Days After Second Product Administration) |  | 8254.41 [6882.60 to 9899.64] | 6494.85 [4097.53 to 10294.75] | 7565.28 [6279.67 to 9114.09]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after each study injection. Unsolicited AEs were recorded from receipt of the first study injection through the visit scheduled 4 weeks after each study injection. At other time periods between injections and when greater than 4 weeks after the last injection, only serious AEs, influenza or influenza-like illness (ILI) and new chronic medical conditions that required ongoing medical management were recorded through the last study visit.
Description: The overall Arms/Groups summarize AEs collected after each product administration separately and grouped by the study product and dose. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity. Influenza/ILI were collected separately and not included as AE.
Arm/Group | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years | Overall Group 2: H10ssF-6473 (60 mcg)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/14 | 0/8 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/14 | 0/8 | 0/22
Other Adverse Events (participants affected / at risk) | 2/3 | 13/14 | 7/8 | 20/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: H10ssF-6473 (20 mcg), Ages 18-50 Years (N=3) | Group 2A: H10ssF-6473 (60 mcg), Ages 18-50 Years (N=14) | Group 2B: H10ssF-6473 (60 mcg), Ages 55-70 Years (N=8) | Overall Group 2: H10ssF-6473 (60 mcg) (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 2
Paronychia (Infections and infestations) | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1
Citrate toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Administration site pain (General disorders) | 0 | 5 | 3 | 8
Administration site swelling (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 1 | 5 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 4
Headache (Nervous system disorders) | 0 | 1 | 2 | 3
Chills (General disorders) | 0 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 — Joint Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT04579250/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT04579250/ICF_000.pdf